CLINICAL TRIAL: NCT04900857
Title: Comparison of Vibration Applied to the Trigger Point and Dry Needle in Acute Myofascial Pain Syndrome: a Prospective Randomized Controlled Research
Brief Title: Comparison of Vibration and Dry Needle in Trigger Point Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IstPMRTRH-MP
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Myofascial Pain Syndrome; Trigger Point Pain, Myofascial
Keywords: Myofascial Pain Syndrome; Trigger Point; Dry Needling; Vibration
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling treatment group (Active Comparator): Dry needling treatment group will be treated with acupuncture needles (0.25x25 mm Hua Long Brand).In this group, one active trigger point area in the trapezius muscle was precisely determined and marked with a permanent pen, and dry needling treatment was applied to that area with disposable acupuncture needles in a single session. the trigger point was palpated. From the center, the needle tip was inserted perpendicular to the skin quickly into the subcutaneous tissue and inserted into the muscle with the needle tip until it found the trigger point in the muscle band. Local twitch responses (LTRs) were similar to Hong's rapid entry and exit technique. It was obtained by inserting a large number of rapid needles in and out of. The needle was not removed from that area for the maximum stimulation time of 1 minute to 3 minutes after a local twitch response was obtained.
  Interventions: Other: Dry needle
- Localized vibration treatment group (Experimental): The tight band in the muscle was determined by palpation, and the location of the most painful points (the middle of the most vertical fibers of the upper part of the trapezius muscle) in the muscle tension band was digitally determined. It was determined with a permanent marker. The skin was cleaned with a suitable antiseptic agent. Localized vibration therapy was applied for 20 minutes with a vibration frequency of 110 Hz and an amplitude of 5.57 mm using a vibrator device. Vibration therapy was applied to our patients by attaching an apparatus with a small area of 1 cm2 to the skin on the trigger point in the trapezius muscle and fixed with medium pressure. We applied a total of 3 sessions every other day in hospital conditions by a single practitioner to all patients.
  Interventions: Device: Localize vibration

INTERVENTIONS:
Other: Dry needle — Local twitch responses (LTRs) were obtained by multiple rapid insertions of the needle in and out of the point, similar to Hong's rapid-entry and rapid exit technique. Hong 1994). The needle was not removed from that site for the maximum stimulation time of 1 minute to 3 minutes after a local twitch response was obtained.
  Arms: Dry needling treatment group
Device: Localize vibration — the vibration was applied with 110 Hz and 5.57 mm amplitude.
  Arms: Localized vibration treatment group

SUMMARY:
The aim of this study is to compare the effects of localized vibration and dry needling applied to the trigger point in the individuals with acute myofascial pain syndrome.Pressure pain threshold (PPT) was used for the primary outcome measure of the study, and pain intensity, pain tolerance and short form (SF-36) were used for secondary outcome measures.

DETAILED DESCRIPTION:
The patients were divided into two groups as dry needling and localized vibration using the permuted block randomization method. The study was completed with 20 (17 women, 3 men) in the dry needling group and 20 in localized vibration (15 women, 5 men). In both applications, a total of 3 sessions were made to the patients at 1-day intervals.Patients' age, gender, duration of pain, localization, presence of additional disease, drug use were questioned and recorded. Pressure pain threshold (PPT) was used for the primary outcome measure of the study, and pain intensity, pain tolerance and short form (SF-36) were used for secondary outcome measures. All evaluation criteria except SF-36 were made before, immediately after and 1 day after each session, 1 week after the last session. SF-36 was evaluated before the 1st session treatment, after the 3rd session treatment and 1 week after the 3rd session treatment.

ELIGIBILITY:
Inclusion Criteria:

* At least one active myofascial trigger point in the upper trapezius muscle
* Symptoms lasting 1 day to 2 weeks
* Cases who did not receive any physical therapy or medication to relieve pain

Exclusion Criteria:

* Sensory defect in the area to be treated with vibration
* Active inflammatory, rheumatological or infectious disease
* Peripheral nerve lesions such as polyneuropathy, radiculopathy
* Having a cardiac disorder (rhythm / conduction disorder, cardiac pacemaker, ischemic heart disease)
* Diagnosis of fibromyalgia or other common musculoskeletal pain syndromes with an intact skin surface in the area to be vibrated
* Patients with a history of panic attacks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Pressure pain threshold | Change from baseline pressure pain threshold score at immediately after, 1 day after and 1 week after the last session
  The test determines the amount of pressure over a given area in which a steadily increasing nonpainful pressure stimulus turns into a painful pressure sensation

SECONDARY OUTCOMES:
Visual analog scale | Change from baseline VAS score at immediately after, 1 day after and 1 week after the last session
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured.
  The patients were asked to score between 0 and 10 for the severity of their pain. It was said that 0 on the scale means no pain, 10 means unbearable pain.
Pain tolerance | Change from baseline Pain tolerance score at immediately after, 1 day after and 1 week after the last session
  Using an algometer (WAGNER-FPK20), a pressure of 2.5 kg /cm2 will be applied to the trigger point and patients will be asked to measure their pain with VAS after pressure application. The severity of the pain felt by the patients after the application of pressure will be measured by VAS. The patients were asked to score between 0 and 10 for the severity of their pain. It was said that 0 on the scale means no pain, 10 means unbearable pain.
Short Form 36 (SF-36) | Change from baseline Short Form 36 score at immediately after the 3rd session and 1 week after the treatment
  The scale consists of 36 items and these provide the measurement of 8 dimensions; physical function (10 items), social function (2 items), role limitations due to physical functions (4 items), role limitations due to emotional problems (3 items), mental health (5 items), energy / vitality (4 items), pain (2 items) and general perception of health (5 items).

CONTACTS AND LOCATIONS:
Overall Officials: Nurdan Paker, Prof, Study Chair — Istanbul Physical Medicine Rehabilitation Training & Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training & Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duenas L, Zamora T, Lluch E, Artacho-Ramirez MA, Mayoral O, Balasch S, Balasch-Bernat M. The effect of vibration therapy on neck myofascial trigger points: A randomized controlled pilot study. Clin Biomech (Bristol). 2020 Aug;78:105071. doi: 10.1016/j.clinbiomech.2020.105071. Epub 2020 Jun 3. PMID 32521284
- [Background] Hong CZ. Lidocaine injection versus dry needling to myofascial trigger point. The importance of the local twitch response. Am J Phys Med Rehabil. 1994 Jul-Aug;73(4):256-63. doi: 10.1097/00002060-199407000-00006. PMID 8043247
- [Background] Issurin VB. Vibrations and their applications in sport. A review. J Sports Med Phys Fitness. 2005 Sep;45(3):324-36. PMID 16230984
- [Background] Kalichman L, Vulfsons S. Dry needling in the management of musculoskeletal pain. J Am Board Fam Med. 2010 Sep-Oct;23(5):640-6. doi: 10.3122/jabfm.2010.05.090296. PMID 20823359